CLINICAL TRIAL: NCT00213408
Title: Catheter Ablation as the First Line Therapy for Symptomatic Typical Atrial Flutter: A Multicenter Randomized Study of Cost/Effectiveness
Brief Title: Catheter Ablation as the First Line Therapy for Typical Atrial Flutter
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: end of the follow-up period
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1999/026/HP
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Atrial Flutter
Keywords: Arrhythmia; atrial flutter; catheter ablation
MeSH Terms: conditions — Atrial Flutter; Arrhythmias, Cardiac

INTERVENTIONS:
Procedure: Radiofrequency catheter ablation of typical atrial flutter

SUMMARY:
Catheter ablation of typical atrial flutter is a well established technique with a high acute success rate and very low complication and recurrence rates. It has also been shown that ablation of recurrent symptomatic typical atrial flutter led to a clear improvement in quality of life. We sought to evaluate the cost/effectiveness of catheter ablation as the first line therapy in patient suffering from their first symptomatic typical atrial flutter episode. This study is a multicenter trial in which patients with a first symptomatic episode of typical atrial flutter are randomized to undergo ablation or to receive antiarrhythmic drugs after electrical cardioversion. Clinical examination, quality of life questionnaires,12 leads ECG and 24-hour Holter monitoring are performed at 1, 3, 6 and 12 months following randomization.The primary end-point is the absence of recurrence of typical atrial flutter at - and 12 months of follow up. The secondary end points are the cost and the cost/effectiveness ratio of these two approaches.

ELIGIBILITY:
Inclusion Criteria:

* first episode of symptomatic typical atrial flutter
* > 18 years old

Exclusion Criteria:

* Prior antiarrhythmic drug treatment for atrial flutter
* History of cavotricuspid isthmus ablation
* Pregnancy
* Hyperthyroidism
* contraindication for anticoagulant therapy
* Life expectancy < 1 year
* contraindication to catheter ablation or to electrical cardioversion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2001-06; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Absence of typical atrial flutter recurrence at 6 and 12 months

SECONDARY OUTCOMES:
Cost/effectiveness ratio at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: frederic Anselme, MD, PhD, Principal Investigator — Service de Cardiologie, Rouen University Hospital
Locations (1):
- CHU de Rouen, Rouen, Seine Maritime, France